CLINICAL TRIAL: NCT07021547
Title: A Single- and Multiple-Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of LY3867070 in Healthy Participants
Brief Title: A Study of LY3867070 in Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 18873; J5H-MC-KVAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-05-21; First posted 2025-06-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Parts A, B, and C are parallel. Part D is open-label fixed-sequence. Part E is crossover.
Who Masked: Participant, Investigator
Masking Description: Part D will be open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3867070 (Part A) (Experimental): Single-Ascending Dose of LY3867070 administered orally
  Interventions: Drug: LY3867070
- LY3867070 (Part B) (Experimental): Multiple-Ascending Doses of LY3867070 administered orally
  Interventions: Drug: LY3867070
- LY3867070 (Part C) (Experimental): Multiple Doses of LY3867070 administered orally
  Interventions: Drug: LY3867070
- Placebo (Parts A-C) (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo
- LY3867070 (Part D) (Experimental): Drug-Drug Interaction (DDI) administered orally
  Interventions: Drug: LY3867070
- LY3867070 (Optional Part E) (Experimental): LY3867070 administered orally
  Interventions: Drug: LY3867070

INTERVENTIONS:
Drug: LY3867070 — Administered orally
  Arms: LY3867070 (Optional Part E); LY3867070 (Part A); LY3867070 (Part B); LY3867070 (Part C); LY3867070 (Part D)
Drug: Placebo — Administered orally
  Arms: Placebo (Parts A-C)

SUMMARY:
The purpose of this study is to evaluate how well LY3867070 is tolerated and what side effects may occur in healthy participants. The study drug will be administered orally. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation
* Part C of the study includes only Japanese and Chinese participants
* Have a body weight greater than or equal to 45 kilogram (kg) and also body mass index 18 to 32 kilogram per square meter (kg/m²) inclusive

Exclusion Criteria:

* Have a history or presence of multiple or severe allergies, anaphylactic reaction to prescription or nonprescription drugs, or history of significant atopy
* Have a significant history or current thyroid disease
* Have a significant history of or current psychiatric disorders, rheumatologic, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (such as Cushing syndrome and hyperaldosteronism), hematological, or neurological disorders
* Are smokers (including electronic cigarettes) within 6 months prior to screening and unwilling to refrain from smoking for the duration of the study.
* Unwilling to undergo skin biopsies (for Part B only)
* Are unwilling to have body hair cut or shaved in cases where hair, in the investigator's opinion, could interfere with noninvasive skin patch

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Approximately Week 7
  A summary of TEAEs regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Approximately Week 7
  A summary of SAEs regardless of causality, will be reported in the Reported Adverse Events module
Number of Participants with One or More Adverse Event(s) (AEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to Approximately Week 7
  A summary of AEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3867070 | Baseline up to Approximately Week 7
  PK: AUC of LY3867070
PK: Maximum Concentration (Cmax) of LY3867070 | Baseline up to Approximately Week 7
  PK: Cmax of LY3867070
Part B Pharmacodynamic (PD): Change from Baseline in Gene Expression | Baseline up to Approximately Week 6
  PD: Change from Baseline in Gene Expression

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Fortrea Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No